CLINICAL TRIAL: NCT06234969
Title: A Mechanistic Trial of the Neurobiology of Extinction Learning and Intraparietal Sulcus Stimulation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Basic Science
Other Study IDs: 849571
Record Dates: First submitted 2024-01-22; First posted 2024-01-31 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Posttraumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Continuous theta burst stimulation to the intraparietal sulcus (Experimental): Continuous theta burst stimulation will be delivered to the individually targeted intraparietal sulcus site at 100% RMT.
  Interventions: Device: Continuous Theta Burst Stimulation to the Intraparietal Sulcus
- Sham continuous theta burst stimulation (Placebo Comparator): We will use the coil's electric stimulation functionality that allows for the delivery of a brief electric pulse to the scalp simultaneous to the pulse to mimic actual stimulation.
  Interventions: Device: Sham Continuous Theta Burst Stimulation

INTERVENTIONS:
Device: Continuous Theta Burst Stimulation to the Intraparietal Sulcus — Continuous Theta Burst Stimulation delivered to the Intraparietal Sulcus
  Arms: Continuous theta burst stimulation to the intraparietal sulcus
Device: Sham Continuous Theta Burst Stimulation — Sham Continuous Theta Burst Stimulation
  Arms: Sham continuous theta burst stimulation

SUMMARY:
This study will be the first of its kind to explore the impact of continuous theta burst stimulation (cTBS) to the intraparietal sulcus (IPS) on arousal symptoms among patients with posttraumatic stress disorder (PTSD). The investigators will demonstrate that IPS cTBS results in significant reduction in arousal (measured by startle response) compared to sham cTBS, that IPS cTBS interacts with extinction training to further improve arousal, and that there is a dose/response effect of cTBS on arousal. The investigators will also demonstrate that IPS cTBS significantly improves retention of extinction learning, the experimental analogue of exposure therapy.

DETAILED DESCRIPTION:
Posttraumatic stress disorder (PTSD) is associated with alterations in arousal that do not respond well to evidence-based practices. Patients with PTSD tend to fall into one of two groups in extinction training (and in exposure therapy): 1) over-engagers, where arousal is too high; and 2) under-engagers, where patients are so worried about becoming upset that they distract themselves from the task (which prevents learning). In this mechanistic clinical trial, the investigators will evaluate a strategy to augment extinction training with neuromodulation to reduce arousal and improve extinction retention. Augmenting extinction training with continuous theta burst stimulation (cTBS, a type of transcranial magnetic stimulation) delivered to the intraparietal sulcus (IPS) may lead to targeted reductions in arousal. The investigative team has shown that the IPS is a "connectivity hub" for arousal and that stimulating this region with TMS can reduce excessive arousal in healthy people. The goal for this R01 is to evaluate the main effects of IPS cTBS (versus sham cTBS, a between-subject comparison) and its interaction with extinction training (vs. neutral training) on arousal among patients with PTSD. The investigators hypothesize that reducing parietal hyperexcitability will help patients with PTSD to modulate arousal during extinction training-enough arousal to ensure that they can benefit, but not too much arousal which prevents learning. These results could translate into future opportunities for novel therapeutic targets among patients with PTSD. The specific aims are as follows: Aim 1: To evaluate the optimal dose of IPS cTBS. H1: Attenuation of startle for IPS cTBS vs. sham cTBS will plateau at 1200 pulses, the anticipated optimal cumulative dose. Aim 2: To compare the main effect of IPS cTBS and its interaction with extinction training on arousal (measured by startle response). Using a two (between group: sham vs. IPS cTBS) x 2 (within group: extinction training vs. control/neutral training) randomized controlled design among patients with PTSD (N = 120), the investigators will examine the potential benefit of cTBS and extinction training on reduction in arousal. H2a: IPS cTBS will result in greater reduction in arousal compared to sham cTBS. H2b: Participants who receive IPS cTBS will have a significantly lower difference in retention of extinction learning vs. control/neutral training (indicative of greater retention of extinction learning) compared to participants who receive sham cTBS. Secondary: The investigators will test analogous hypotheses on subjective outcomes and on cognitive outcomes and the investigators hypothesize similar directions of effects. Aim 3: To evaluate neural mechanisms of action of IPS cTBS + extinction training. Participants will complete a resting state fMRI scan on tests of retention of learning experimental visits to evaluate neural changes from training. H3: The investigators will observe attenuated activation (relative to pre-test) of the IPS for participants who received IPS cTBS compared to those who received sham cTBS.

ELIGIBILITY:
Inclusion Criteria:

* Adult aged 18-60
* Meets Diagnostic and Statistical Manual of Mental Disorders (DSM-5) criteria for PTSD according to the Clinician-Administered PTSD Scale for DSM-5
* No metal implants

Exclusion Criteria:

* Pregnancy
* Seizure disorder or epilepsy
* Increased risk of seizure
* Non-English speaking
* Any medical condition that increases risk for fMRI or cTBS
* Medical implant
* Hearing loss sufficient to interfere with startle
* Claustrophobia
* Recent medication or therapy changes (in the past 8 weeks)
* Current severe substance use disorder

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-04-29 (Actual); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
Electromyography startle response | Days 4, 5, 34 and 35
  Startle will be recorded from the left orbicularis oculi at 2000 Hz.

SECONDARY OUTCOMES:
Subjective Units of Distress (SUDS) | Days 4, 5, 34 and 35
  We will assess SUDS using the prompt "On a scale from 0 - 10, how distressed does this recording make you?"
Negative outcome expectancy | Days 4, 5, 34 and 35
  On a scale from 0 ("certain no negative outcome") to 10 ("certain negative outcome"), how certain are you that the negative outcome will happen as you listen this script?
fMRI | Days 2, 5, and 35
  We will collect resting state functional connectivity.

CONTACTS AND LOCATIONS:
Overall Officials: Lily A Brown, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- Center for the Treatment and Study of Anxiety, University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share data through the NIMH Data Archive using only de-identified data connected through the global unique identifier (GUID).
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be entered into the NIMH Data Archive every 6 months.
URL: https://nda.nih.gov/